CLINICAL TRIAL: NCT01445847
Title: Effect of Intravenous Lidocaine on the Incidence of Post-extubation Laryngospasm: A Randomised Controlled Trial
Brief Title: The Effect of Intravenous Lidocaine on Post-extubation Laryngospasm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient Safety Concerns
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Khalid Ibrahim Aljonaieh, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: E-11-491
Record Dates: First submitted 2011-09-29; First posted 2011-10-04 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Laryngospasm
Keywords: Laryngospasm; Lidocaine
MeSH Terms: conditions — Laryngismus | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine 1% was prepared in 10 mL syringe= 10 mg/mL, dosage was 1mg/kg, one bolus or 10 mL/kg, with range of 2mg could be added or missed. The maximum dose is 100 mg for patients with weight of more than 100
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Normal saline was prepared in 10 mL syringe, dosage was 1 mL/10 kg.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine — 1 mg/kg or 1 mL/10 kg prior to extubation period. Injection of Lidocaine will be immediately when inhalational agent (Desflurane) is discontinued.
  Other Names: Xylocaine
  Arms: Lidocaine
Other: Placebo — 1 mL/10 kg prior to extubation period. Injection of placebo will be immediately when inhalational agent (Desflurane) is discontinued.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
In the literature, we found no randomized clinical trials addressing the using of IV lidocaine as prophylaxis for postoperative laryngospasm among adults.

The aim of this study was to assess the effects of IV lidocaine on the incidence of postoperative laryngospasm of adults patients.

DETAILED DESCRIPTION:
During anesthesia practice, one of the common complications of airway management is laryngospasm. The etiology of laryngospasm is unknown but may be due to insufficient depth of anesthesia during tracheal intubation, light plane of anesthesia during tracheal extubation, pain, or presence of airway irritant like laryngoscope blade, irritated volatile agent, suction catheter, surgical debris, mucus, blood, or other foreign body. Laryngospasm occurs in both genders and all ages. Incidence of laryngospasm was reported to the Australian incident monitoring study (AIMS) was 5% with of 22% of them without an attributable cause.

Currently, there is no proven prophylaxis for laryngospasm and the known treatments of laryngospasm are used post-occurrence. However, elimination of factors that lead to laryngospasm is the most indispensable item for reduction of its incidence.

Intravenous (IV) lidocaine interrupts nerve conduction by blocking sodium channels. Recent meta-analysis study showed that IV lidocaine was able to prevent laryngospasm in children. However, in the literature, we found no randomized clinical trials addressing the using of IV lidocaine as prophylaxis for postoperative laryngospasm among adults.

The aim of this study was to assess the effects of IV lidocaine on the incidence of postoperative laryngospasm of adults patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia score are I or II
* Undergo for laparoscopic cholecystectomy

Exclusion Criteria:

* Patient's refusal
* History of upper respiratory tract infection (URTI) within 2 weeks
* Persistent type of hyper-reactive airway or asthma
* History of airway surgery
* History of gastro-esophageal reflex disease (GERD)
* Currently receiving sedating or analgesic medication
* Currently receiving the following medications:

  * Fluvoxamine
  * Erythromycin and Itraconazole
  * β -blocker or Cimetidine
* History of Lidocaine Allergy
* History of epilepsy disorder
* Pregnant or breastfeeding women
* History of Heavy Smoking ( a smoker with a daily cigarettes consumption of more than 20 pieces
* History of increased salivation by a disease or medication
* History of difficult intubation
* Two or more attempts of intubation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khalid I Aljonaieh, Lecturer, Principal Investigator — King Saud University
Locations (1):
- College of Medicine - King Saud University Medical City, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- See also: King Saud University — http://ksu.edu.sa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted at King Khalid University Hospital, King Saud University, Riyadh, Saudi Arabia at Jan 20, 2012. Recruitment was done at Their wards within 24 hours prior to the operation
Pre-assignment Details: Patients were able to refuse to participate before anesthesia induction start. Therefore, patients may excluded from the study due to that reason and we decided to start assignment to groups randomly when anesthesia is induced to the patient.
Groups:
- Lidocaine: Lidocaine group received 1 mL/10 kg (or 1 mg/kg) bolus once inhalational gas (Desflurane) is discontinued
- Placebo: Placebo group received 1 ml per 10 kg bolus once inhalational gas (Desflurane) is discontinued
Period: Overall Study
Arm/Group | Lidocaine | Placebo
Started | 50 | 50
Completed | 36 | 36
Not Completed | 14 | 14
Not completed — Protocol Violation | 13 | 14
Not completed — Missed Data | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo group received 1 mL/10 kg bolus once inhalational gas (Desflurane) is discontinued
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.61 (8.73) | 39.39 (10.84) | 38.01 (10.51868595)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Laryngospasm Postoperatively
Description: There were 4 scores of laryngospasm:
  0 = No Laryngospasm
  1. = Stridor or partial laryngospasm
  2. = Complete Laryngospasm
  3. = Cyanosis
Time Frame: within first 15 minutes post-dose
Population: Trial was terminated by data monitoring committee due to safety concerns
Measure: Number; unit: participants
Groups:
- Lidocaine: Lidocaine group received 1 mg per kg (1mL per 10kg) bolus once inhalational gas (Desflurane) is discontinued
- Placebo: Placebo group received 1 ml per 10 kg (0.2 mL per 2 kg) bolus once inhalational gas (Desflurane) is discontinued
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 36 | 36
participants | 0 | 7
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; We used incidence reported to AIMS study to calculate the sample size of this study. We set the null hypothesis as (percentage point of laryngospasm incidence in placebo group (µ1) - percentage point of laryngospasm incidence in Lidocaine group (µ2) = 0), with alternative hypothesis is (µ1 > µ2) by 5% was analyzed by comparison of two proportions. A sample size of 380 patients (190 per group) was adequate to detect a 5-percentage point difference in the incidence with 80% power and p = 0.05; Test type: Superiority or Other; p < 0.05, Comparison of proportions; Percentage = 5, 95% CI 2-sided [1.7 to 9.1]

ADVERSE EVENTS:
Time Frame: within 4 months
Groups:
- Lidocaine: Lidocaine group received 1 ml/10 kg (or 1mg/kg) bolus once inhalational gas (Desflurane) is discontinued
Arm/Group | Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 7/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=36) | Placebo (N=36)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)

LIMITATIONS AND CAVEATS:
Early termination of the trial led to small numbers of subjects that received allocated intervention, (i.e., 99 total participants).

Additionally, protocol violation led to reduce the analyze subjects to 36 for each group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes